CLINICAL TRIAL: NCT06849713
Title: A Phase 2 Study of Zanubrutinib, Obinutuzumab, and Sonrotoclax in Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Zanubrutinib, Obinutuzumab, and Sonrotoclax in Previously Untreated Patients With CLL or SLL
Acronym: BOSon
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Principal Investigator, Jacob Soumerai, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-007
Record Dates: First submitted 2025-02-12; First posted 2025-02-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma (SLL)
Keywords: CLL; SLL; untreated
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib, obinutuzumab, and sonrotoclax (Experimental): Zanubrutinib will be taken orally twice daily on days 1-28 of each cycle.
  Sonrotoclax will be taken orally once daily on days 1-28 starting cycle 3 day 1.
  Obinutuzumab will be given into the vein (by intravenous infusion) at the following timepoints: Days 1, 8, and 15 of cycle 1, Day 2 of cycle 1, and Day 1 of cycles 2 through 6.
  The total regimen treatment duration depends on early MRD response kinetics (ΔMRD400). The total regimen treatment duration will be 10 cycles for patients who achieve ΔMRD400 and 24 cycles for patients who do not achieve ΔMRD400 (including the 2-month zanubrutinib/obinutuzumab lead-in).
  Drug diaries will be provided to participants to document information about zanubrutinib and sonrotoclax.
  Interventions: Drug: Zanubrutinib; Drug: Sonrotoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Zanubrutinib — Bruton's Tyrosine Kinase (BTK) inhibitor
  Other Names: BGB-3111
Drug: Sonrotoclax — B-cell lymphoma 2 (BCL2) protein inhibitor
  Other Names: BGB-11417
Drug: Obinutuzumab — Anti-CD20 monoclonal antibody

SUMMARY:
The purpose of this study is to determine the proportion of participants who achieve undetectable measurable residual disease (uMRD) in previously untreated chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
This is a multicenter phase II study evaluating zanubrutinib, obinutuzumab, and sonrotoclax in previously untreated patients with CLL or SLL.

Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved sonrotoclax as a treatment for any disease.

The U.S. Food and Drug Administration (FDA) has approved zanubrutinib and obinutuzumab as a treatment option for your disease.

The combination of zanubrutinib, obinutuzumab, and sonrotoclax (BOSon regimen) is not an approved regimen for CLL or SLL and is investigational in this study.

The duration of the protocol therapy will depend on participant's individual response, with a longer course of therapy for participants with a lower response, and a shorter course of therapy for those with a faster response. After removal from the protocol therapy, participants will be followed for up to 2 years after the final patient is enrolled.

It is expected that about 40 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have CLL or SLL (WHO criteria).
* Participant must require treatment according to iwCLL guidelines.
* Participants must have no prior systemic therapy for CLL or SLL, except:

  * Prior local radiation for symptomatic disease is permitted.
  * Short course systemic corticosteroids is permissible for disease control, improvement of performance status, or non-cancer indication. However, duration of steroid course must be ≤14 days with maximum daily dose of ≤100 mg prednisone, ≤20 mg dexamethasone, or equivalent, and must be discontinued prior to study treatment (last dose may be administered up until the morning of / prior to study treatment). Inhaled steroids, topical steroids, and replacement / stress corticosteroids are permitted independent of above rules. In cases of autoimmune complications of CLL (e.g., ITP or AIHA), steroid usage is permitted.
* Age ≥18 years.
* ECOG performance status of 0, 1 or 2.
* Participants must meet the following organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/µL without growth factor support (filgrastim within 5 days or PEGfilgrastim within 10 days of test), unless clearly due to disease under study (per investigator)
  * platelets ≥75,000/µL, or ≥20,000/µL if clearly due to disease under study (per investigator)
  * total bilirubin ≤2 x institutional upper limit of normal (ULN), or ≤3 x institutional ULN if due to Gilbert's syndrome, or with PI approval if clearly due to disease under study
  * AST(SGOT)/ALT(SGPT) ≤2.5 x × institutional ULN
  * CrCl or GFR ≥30 mL/min as estimated by the Cockcroft-Gault equation, the CKD-EPI equation, or as measured by 24-hour urine collection
* For females of childbearing potential, a serum pregnancy test must be negative within screening period.
* For female patients of childbearing potential: agreement to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) or remain abstinent (refrain from heterosexual intercourse) during the treatment period and to continue its use for ≥ 30 days after the last dose of zanubrutinib or ≥ 90 days after the last dose of sonrotoclax, and for ≥18 months fter the last dose of obinutuzumab (whicher is later).

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Hormonal contraceptive methods must be supplemented by a barrier method.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men with a female partner of childbearing potential or a pregnant female partner: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom in addition to 1 of the highly effective methods of contraception listed below, from the time of taking the first dose of study drug , during the treatment period and to continue its use for ≥ 30 days after the last dose of zanubrutinib or ≥ 90 days after the last dose of sonrotoclax, and for ≥18 months fter the last dose of obinutuzumab (whicher is later).

  --The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Willingness to not donate or bank sperm or oocytes during the entire study treatment period and after treatment discontinuation for for ≥ 30 days after the last dose of zanubrutinib or ≥ 90 days after the last dose of sonrotoclax, and for ≥18 months fter the last dose of obinutuzumab (whicher is later).
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)

Exclusion Criteria:

* Known histologic transformation from CLL or SLL to an aggressive lymphoma (i.e., Richter's transformation).
* Known central nervous system involvement with CLL or SLL.
* Other diagnosis of active malignancy or systemic therapy within 2 years of study treatment. Note: An active malignancy or systemic therapy within 2 years for another malignancy, whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Also, local/regional therapy with curative intent such as surgical resection or localized radiation at any timepoint is permitted.
* Any uncontrolled illness that in the opinion of the investigator would preclude administration of study therapy (e.g., significant active infections, hypertension, angina, arrhythmias, pulmonary disease, or autoimmune dysfunction).
* Congestive heart failure, New York Heart Association III/IV. Unstable angina within 3 months before screening, myocardial infarction within 6 months before screening. History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes). Heart rate-corrected QT interval > 480 milliseconds based on Fridericia's formula corrected for bundle branch block as appropriate. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place.
* Receipt of a live-virus vaccine within 28 days prior to initiation of study treatment or need for live-virus vaccine at any time during study treatment.
* Active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds).
* Known bleeding diathesis. History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention.
* Prior major surgical procedure within 4 weeks of study, or anticipation of need for a major surgical procedure during the course of the study.
* Known CNS hemorrhage or stroke within 6 months of the study.
* History of progressive multifocal leukoencephalopathy.
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection.

  * Patients with a history of HIV infection that is well controlled on antiretroviral therapy are eligible if all of the following criteria are met: (1) undetectable HIV viral load by standard clinical assay AND (2) CD4+ T cell count of >/=200 cells/microliter). NOTE: Many HIV regimens are excluded based on drug interactions, and concomitant antiretroviral therapy must be acceptable per protocol.
  * Participants with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable, and if the participant is willing to take appropriate anti-viral prophylaxis as indicated and HBV DNA monitoring on study.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.

Known condition or other clinical situation resulting in inability to swallow oral medications, or that would impair absorption of oral medications.

* Participant in a separate investigational therapeutic trial unless authorized by the PI.
* Concurrent therapy with, or administration within 5 half-lives 14 days prior to the first dose of study drug (whichever is shorter), with moderate or strong inhibitors or inducers of CYP3A.
* Concomitant use of warfarin or warfarin derivatives.
* Concomitant use of dual antiplatelet therapy.
* Prior systemic therapy for CLL or SLL, except for localized radiation or corticosteroids as per 3.1.3.
* Prior anti-CD20 monoclonal antibody therapy for any indication (malignant or non-malignant).
* Participants with a contraindication to obinutuzumab based on known hypersensitivity (IgE-mediated) reaction to obinutuzumab or to any of its excipients. Hypersensitivity to zanubrutinib or sonrotoclax.
* Consumption of one or more of the following within 3 days prior to the first dose of study drug: grapefruit or grapefruit products, Seville oranges including marmalade containing Seville oranges, or Star fruit (carambola).
* Known psychiatric illness or social situation that would interfere with study adherence.
* Pregnant women are excluded from this study given potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued prior to the first dose of study drug if the mother is treated.
* Uncontrolled autoimmune anemia and/or autoimmune thrombocytopenia (eg, idiopathic thrombocytopenia purpura), e.g., with need for ongoing corticosteroid treatment (see 3.2.24).
* Requires ongoing need for corticosteroid treatment. NOTE: Systemic corticosteroids must be fully tapered off/stopped before first study drug.
* Uncontrolled hypertension at Screening, defined as systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mmHg by ≥ 2 consecutive measurements. In patients NOT meeting these parameters for uncontrolled hypertension, repeat blood pressure measurement is NOT required for eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Undetectable MRD (uMRD) at Best Response | Day 1 to 2 years after final patient enrolled
  The proportion of patients achieving undetectable MRD in peripheral blood using the ClonoSEQ assay (cutoff, <10-5). The number of responses will be reported with a proportion with 95% exact binomial confidence interval.
Proportion of Participants with Tumor Lysis Syndrome (TLS) Laboratory Abnormalities Requiring Intervention | Day 1 to completion date of sonrotoclax ramp-up
  The proportion of participants who have 1 or more TLS laboratory abnormalities requiring intervention on a ramp-up date with normal pre-dose TLS parameters and ALC <25,000/µl during the sonrotoclax ramp-up. The number of responses will be reported with a proportion with 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Frequency of uMRD at Best Response | Day 1 to 2 years after final patient enrolled
  The proportion of patients achieving uMRD in both peripheral blood (PB) and bone marrow (BM) by ClonoSEQ (cutoff, <10-5).
Rate of uMRD after 10 and 24 cycles | Day 1 to end of 10 cycles and end of 24 cycles
  The proportion of patients achieving uMRD in both PB and BM by ClonoSEQ (cutoff, <10-5) after 10 and 24 cycles.
Rate of Complete Response (CR) or CR with Incomplete Marrow Recovery (CRi), or Partial Response (PR) | Day 1 to 2 years after final patient enrolled
  Patients will have their response classified per the 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines.
Progression-free survival (PFS), Overall Survival (OS), MRD4-Free Survival, and MRD5-free survival | Day 1 to first documented disease progression or date of death from any cause, assessed for 2 year after final patient enrolled
  PFS is the time from treatment start to the earlier of progression or death due to any cause. OS is the time from treatment start to death due to any cause. MRD4-Free Survival is the time from treatment start to the earlier of detectable MRD ≥10-4 by immunosequencing (Adaptive ClonoSEQ assay), progression, or death due to any cause. MRD5-Free Survival the time from treatment start to the earlier of detectable MRD ≥10-5 by immunosequencing (Adaptive ClonoSEQ assay), progression, or death due to any cause. Time-to-event endpoints will be evaluated using the Kaplan-Meier method. Survival distributions may be described as medians or 1- and 2-year probabilities with 95% confidence intervals. Uni- and multi-variable Cox regressions may also be performed and will be summarized with hazard ratios, 95% confidence intervals, and Wald p-values.
Proportion of Participants Without TLS-related Laboratories Requiring Clinical Intervention | Day 1 to end of Cycle 3 (each cycle is 28 days)
  TLS is defined according to Howard criteria. The nature, frequency, severity, and timing of TLS will be tabulated and summarized descriptively.
Distribution of TLS Risk | Day 1 to end of Cycle 2 (each cycle is 28 days)
  TLS is defined according to Howard criteria. The nature, frequency, severity, and timing of TLS will be tabulated and summarized descriptively.
Incidence and Severity of Treatment-Emergent Adverse Events | Day 1 to 2 years after final patient enrolled
  Patients will have their toxicities graded and reported at every visit according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The nature, frequency, severity, and timing of adverse events will be tabulated and summarized descriptively. The safety analyses will include all participants who received at least one dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Soumerai, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Jacob Soumerai, MD (jsoumerai@mgh.harvard.edu) at 617-724-4000. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation